CLINICAL TRIAL: NCT01165073
Title: Short Term Feeding for Hospitalised Asian Patients With Liver Cirrhosis - a Randomised Trial of Naso-gastric vs Oral Feeding
Brief Title: Short Term Feeding for Asian Patients With Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Dr Sanjiv Mahadeva/ Dr Sharon Tai Mei Ling, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGVOC1
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2010-07

CONDITIONS: CIRRHOSIS
Keywords: Cirrhosis; Malnutrition; Enteral nutrition
MeSH Terms: conditions — Fibrosis; Malnutrition | interventions — Osmolite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naso-gastric tube feeding (Experimental)
  Interventions: Dietary Supplement: Osmolite and B.C.A.A.
- Oral feeding (Active Comparator)
  Interventions: Dietary Supplement: Normal oral intake & supplementation if necessary

INTERVENTIONS:
Dietary Supplement: Osmolite and B.C.A.A. — Feeding inserted into enteral tubes
  Other Names: Enteral supplementation
  Arms: Naso-gastric tube feeding
Dietary Supplement: Normal oral intake & supplementation if necessary — Enteral nutrition
  Other Names: Enteral supplementation
  Arms: Oral feeding

SUMMARY:
The benefits of short-term naso-gastric feeding in patients with advanced cirrhosis remain uncertain. This was a randomised study comparing naso-gastric feeding and oral feeding in Asian patients with cirrhosis who were admitted to hospital for decompensation.

DETAILED DESCRIPTION:
Consecutive patients with decompensated cirrhosis who fitted the inclusion criteria, will be randomised to either naso-gastric or oral feeding. Total feeding will be for 2 weeks only. Following intervention specific nutritional and liver-related parameters will be measured during the 2 weeks and up to 6 weeks later. Comparison between both groups will then be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated cirrhosis of any etiology.

Exclusion Criteria:

* Advanced hepatic encephalopathy,
* Variceal bleeding,
* Hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improvement in Child-Pugh score | Up to 6 weeks
  Change in the Child-Pugh score, assessing liver damage in cirrhosis

SECONDARY OUTCOMES:
Improvement in nutritional parameters | up to 6 weeks
  Improvement in nutritional anthropometry and assessment tool markers after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Mahadeva, MRCP, Study Director — University of Malaya; Mei-Ling S Tai, MRCP, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Cabre E, Gonzalez-Huix F, Abad-Lacruz A, Esteve M, Acero D, Fernandez-Banares F, Xiol X, Gassull MA. Effect of total enteral nutrition on the short-term outcome of severely malnourished cirrhotics. A randomized controlled trial. Gastroenterology. 1990 Mar;98(3):715-20. doi: 10.1016/0016-5085(90)90293-a. PMID 2105256
- [Result] Campillo B, Richardet JP, Bories PN. Enteral nutrition in severely malnourished and anorectic cirrhotic patients in clinical practice. Gastroenterol Clin Biol. 2005 Jun-Jul;29(6-7):645-51. doi: 10.1016/s0399-8320(05)82150-5. PMID 16141996
- [Result] Campillo B, Richardet JP, Scherman E, Bories PN. Evaluation of nutritional practice in hospitalized cirrhotic patients: results of a prospective study. Nutrition. 2003 Jun;19(6):515-21. doi: 10.1016/s0899-9007(02)01071-7. PMID 12781851
- [Result] Kondrup J, Muller MJ. Energy and protein requirements of patients with chronic liver disease. J Hepatol. 1997 Jul;27(1):239-47. doi: 10.1016/s0168-8278(97)80308-x. No abstract available. PMID 9252101
- [Result] Plauth M, Merli M, Kondrup J, Weimann A, Ferenci P, Muller MJ; ESPEN Consensus Group. ESPEN guidelines for nutrition in liver disease and transplantation. Clin Nutr. 1997 Apr;16(2):43-55. doi: 10.1016/s0261-5614(97)80022-2. No abstract available. PMID 16844569
- [Result] Alvares-da-Silva MR, Reverbel da Silveira T. Comparison between handgrip strength, subjective global assessment, and prognostic nutritional index in assessing malnutrition and predicting clinical outcome in cirrhotic outpatients. Nutrition. 2005 Feb;21(2):113-7. doi: 10.1016/j.nut.2004.02.002. PMID 15723736